CLINICAL TRIAL: NCT04890587
Title: A Dose Escalation Tolerance and Pharmacokinetics Study of AL8326 in Advanced Solid Tumor
Brief Title: A Phase I Study of AL8326 in Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Advenchen Laboratories Nanjing Ltd. (Industry)
Responsible Party: Sponsor
Organization: Advenchen Laboratories, LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL8326-CN-001
Record Dates: First submitted 2021-04-26; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Advanced Solid Tumors
Keywords: Maximum tolerated dose; Dose limiting toxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AL8326 (Experimental): Part 1:(closed)Cohort 1 will initiate with AL8326 for single dose and multiple dose (28-Day cycles) . After three subjects have completed the first cycle of therapy without a DLT, additional cohorts may be enrolled sequentially. After the first cohort has completed one full cycle of therapy without a DLT, several additional cohorts will be sequentially for the same 28-day cycles.
  Part 2 :(open)Each subject will receive a dose from Part 1 of this study for continuous 28-Day cycles of therapy.
  Part 3:(open)Cohort 3 will initiate with AL8326(bid), for 28-Day cycles . After three subjects have completed the first cycle of therapy without a DLT, additional cohorts may be enrolled sequentially. After the first cohort has completed one full cycle of therapy without a DLT, two additional cohorts will be sequentially enrolled at decreased dose of AL8326 for the same 28-day cycles.
  Interventions: Drug: AL8326 tablets

INTERVENTIONS:
Drug: AL8326 tablets — Tablet:10mg/tablet; administered orally once daily in part 1 and part 2, administered orally twice daily for continuous 28-Day cycles in part 3.
  Other Names: AL8326

SUMMARY:
1. Main purpose Objective to study the tolerance and safety of single and multiple administration of repeated 28-day cycles of AL8326 in patients with advanced solid tumor, observe the dose limiting toxicity (DLT) and maximum tolerated dose (MTD).
2. Secondary purpose 1) Preliminary analysis of the pharmacokinetic characteristics and efficacy of repeated 28-day cycles of AL8326 tablets in patients with advanced solid tumors; 2) According to the results of phase I tolerance test and pharmacokinetics, appropriate dosage and regimen were recommended for phase II clinical trial;

DETAILED DESCRIPTION:
This is a Phase 1 study to evaluate the safetyand efficacy of 28-day cycles of AL8326 therapy. The study is divided into three parts.

1. Part I To evaluate the dose limiting toxicity (DLT) and general safety during the first 28-day cycle of Al8326 therapy and to evaluate the MTD. It will include a evaluation of 3 subjects per cohort in a 3+3 design in.
2. Part II Subject will receive a dose from Part 1 of this study for continuous 28-Day cycles of therapy.
3. Part III This design adopts 3 + 3 dose de-escalation method for exploration. At the same time, the safety, tolerance and pharmacokinetics were observed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the following advanced solid tumors confirmed by histology or cytology (including but not limited to non-small cell lung cancer, cervical cancer, ovarian cancer, breast cancer, pancreatic cancer, liver cancer, colon cancer, head and neck cancer, prostate cancer, kidney cancer, etc.). Lack of effective standard treatment options; or failure (including disease progression or intolerance) or recurrence after conventional standard treatment.
2. For subject received cytotoxic drugs chemotherapy before, the interval between the end of chemotherapy and the signing of informed consent was at least 4 weeks, and must be recovered from the toxic reaction of previous chemotherapy to ≤ 1 grade (except for hair loss);
3. There must be at least measurable lesions in accordance with RECIST 1.1. If there is only one lesion, the lesion must be confirmed by cytology / histology.
4. Main organ function:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 / L (1500 / mm ^ 3), platelet ≥ 75 × 10 ^ 9 / L or hemoglobin ≥ 9g / dl.
   2. Serum total bilirubin ≤ 2 times the upper limit .
   3. Serum creatinine ≤ 1.5 times the upper limit of normal value or creatinine clearance rate ≥ 50ml / min.
   4. If there is no liver metastasis, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 times of the upper limit, or liver metastasis ≤ 5 times of the upper limit .
   5. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ 50%.
   6. According to the judgment of the investigator, the laboratory examination results and clinical abnormalities that will not affect the safety of the subjects and the completion of the trial can be arranged into the group.
5. ECOG (PS) score was 0,1;
6. Life expectancy ≥ 12 weeks;
7. Age ≥ 18 years old and ≤ 70 years old;
8. There was no malabsorption or other gastrointestinal diseases affecting drug absorption.
9. Female: for female patients with fertility, pregnancy test must be conducted before treatment, and contraceptive method approved by medical department must be adopted during treatment and within 3 months after treatment; serum or urine pregnancy test in screening period must be negative; it must be non lactation period; and；if a female patient is postmenopausal but has not yet reached the postmenopausal state (the duration of menopause is greater than or equal to 12 consecutive months, and there is no other reason except menopause), and has not received sterilization surgery (removal of ovaries and / or uterus), she is considered to be fertile.
10. Male: during surgical sterilization or treatment and within 3 months after the end of the treatment, the contraceptive measures approved by the doctor were adopted;
11. Ability to understand and sign informed consent.

Exclusion Criteria:

1. It is known that it is allergic to drugs with similar chemical structure.
2. Use of drugs or other trial drugs without approval within 30 days before enrollment.
3. The condition of each organ system was as follows：

   1. Patients with previous history of central nervous system metastasis or uncontrollable symptoms of brain metastasis, spinal cord compression and cancerous meningitis within 8 weeks after the first administration. For patients with CNS metastasis or spinal cord compression, if the clinical status is stable and does not need hormone therapy, and the interval between the treatment (including radiotherapy or surgery) before entering the group is more than 4 weeks, they can participate in this trial.
   2. Grade 2 or above hypertension that cannot be controlled by single drug.
   3. Acute myocardial infarction occurred within 6 months.
   4. At present, there are arrhythmias (such as long QT syndrome, unmeasurable or ≥ 480ms of Bazett's corrected QTC).
   5. NYHA cardiac function grade III or IV.
   6. Evidence of severe or uncontrollable systemic disease (e.g., unstable or decompensated respiratory, heart, liver, or kidney disease), as judged by the investigators.
   7. Any unstable systemic disease (including active infection, angina pectoris, liver and kidney or metabolic disease, etc.).
   8. Other (primary) malignancies (except for completely cured cervical carcinoma in situ or basal cell carcinoma or squamous cell skin carcinoma) within five years.
   9. The presence of clinically detectable third space effusion (such as ascites or pleural effusion) requires immediate drainage. Or after treatment, the effusion is not well controlled and continues to increase.
   10. Previous history of definite neurological or mental disorders, such as epilepsy or dementia.
4. The function level of each organ was as follows：

   1. The results of urine protein analysis showed that urine protein was ≥ + +, and 24-hour urine protein was more than 1.0 g.
   2. Coagulation dysfunction: Patients with bleeding tendency (such as active peptic ulcer) or undergoing thrombolytic or anticoagulant therapy; under the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, it is allowed to use low-dose warfarin (1mg oral, once a day) or low-dose aspirin (less than 100mg daily) for preventive purposes.
   3. Patients with arteriovenous thrombosis events within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism.
5. The patients who had been enrolled before who had withdrawn from this study.
6. HIV antibody is positive, or the patient has other acquired or congenital immunodeficiency disease, or has a history of organ transplantation.
7. At the same time, they received any other anti-tumor treatment.
8. The researcher thinks that it is not suitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-17 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | cycle1 (each cycle is 28-days)
  To observe the durability and safety of AL8326 in patients with advanced solid tumor after single and multiple administration, observe the dose limiting toxicity (DLT)and the reversibility of toxicity;
Maximum tolerated dose (MTD) | cycle1 (each cycle is 28-days)
  To observe the durability and safety of AL8326 in patients with advanced solid tumor after single and multiple administration, observe the maximum tolerated dose (MTD)，the relationship between toxicity and dose;

SECONDARY OUTCOMES:
Cmax | cycle1 (each cycle is 28-days)
  The pharmacokinetic characteristics of Al8326 tablets in patients with advanced solid tumor were analyzed;
Tmax | cycle1 (each cycle is 28-days)
  The pharmacokinetic characteristics of Al8326 tablets in patients with advanced solid tumor were analyzed;
AUC0-t | cycle1 (each cycle is 28-days)
  The pharmacokinetic characteristics of Al8326 tablets in patients with advanced solid tumor were analyzed;
AUC0-∞ | cycle1 (each cycle is 28-days)
  The pharmacokinetic characteristics of Al8326 tablets in patients with advanced solid tumor were analyzed;
Vd | cycle1 (each cycle is 28-days)
  The pharmacokinetic characteristics of Al8326 tablets in patients with advanced solid tumor were analyzed;
Ke | cycle1 (each cycle is 28-days)
  The pharmacokinetic characteristics of Al8326 tablets in patients with advanced solid tumor were analyzed;
CL | cycle1 (each cycle is 28-days)
  The pharmacokinetic characteristics of Al8326 tablets in patients with advanced solid tumor were analyzed;
t1/2 | cycle1 (each cycle is 28-days)
  The pharmacokinetic characteristics of Al8326 tablets in patients with advanced solid tumor were analyzed;
Primary antitumor efficiency of AL8326 | Every 3 cycles(each cycle is 28-days)
  Patients with advanced solid tumors and their efficacy in patients with advanced solid tumors were evaluated according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, Principal Investigator — Central organization
Locations (2):
- China (2):
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong